CLINICAL TRIAL: NCT01477268
Title: Determining the Impact of Dementia and Executive Impairment on Antidepressant Treatment Response in Older Persons
Brief Title: Cognitive Correlates of Antidepressant Treatment Response in Elders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Dr. Corinne E. Fischer, St. Michael's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-296
Record Dates: First submitted 2009-06-09; First posted 2011-11-22 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-05

CONDITIONS: Depression
Keywords: antidepressants; depression; zoloft; psychiatry; psychology
MeSH Terms: conditions — Depression | interventions — Sertraline; Antidepressive Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- zoloft (Other): Both arms of the study will include zoloft. However, the treatment response to zoloft will be compared in two different subgroups.
  Interventions: Drug: Zoloft (antidepressant)

INTERVENTIONS:
Drug: Zoloft (antidepressant) — Zoloft 50-200 mg po od x 12 weeks
  Other Names: Sertraline

SUMMARY:
Major depression is a very common health problem affecting older persons. The present standard of treatment is with medications called "antidepressants". Antidepressants have been studied extensively in older persons with normal brain function and have been shown to be effective. However, certain types of brain dysfunction called "executive impairment" (inability to do higher order thinking) may lead to poor treatment outcomes. This study will compare how older depressed people with different levels of executive impairment respond differently to standard antidepressant treatment. Knowing this information will lead to more rational targeting of available treatments, leading to improved treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* above the age of 65,
* speak English fluently,
* experience depression, AND
* not yet on active treatment.

Exclusion Criteria:

* active delirium,
* substance abuse,
* mental illness other than major depression,
* active CNS disease,
* unstable systematic medical disease, OR
* current of past psychotic disorder.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-06; Primary Completion 2009-04 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
depression | June 1, 2007 - June 1, 2008

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Fischer, MD, Principal Investigator — St. Michaels Hospital
Locations (1):
- St Michael's Hospital, Toronto, Ontario, Canada